CLINICAL TRIAL: NCT00393146
Title: A Randomized, Double Blind, Placebo Controlled Study to Investigate the Safety and Tolerability and Clinical Activity of 28 Days of Oral Repeat Dosing With GW856553 at 7.5mg BID in Subjects With Active Rheumatoid Arthritis on Stable Anti-rheumatic Therapy.
Brief Title: A Study To Investigate The Effect Of 28 Days Of Dosing With GW856553 On Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RA3103718
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis; MRI
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW856553 — Study drug

SUMMARY:
This study is designed to look at the safety, tolerability and effectiveness of 28 days of dosing of GW856553 in rheumatoid arthritis patients.

ELIGIBILITY:
Inclusion criteria:

* The subject is male or female ≥ 18 years of age.
* To be eligible, female subjects must have a negative pregnancy test (i.e. serum beta hCG test) and be of:

  1. non-childbearing potential (i.e. physiologically incapable of becoming pregnant). This includes any female who is post-menopausal. For the purposes of this study, post menopausal is defined as being amenorrhoeic for greater than 2 years with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms. Postmenopausal status will be confirmed by serum FSH and oestradiol concentrations at screening. Surgical sterility will be defined as females who have had a hysterectomy and/or bilateral oophorectomy or tubal ligation. OR
  2. childbearing potential and agrees to commit to one of the protocol-approved methods of contraception as detailed in Section 7.1.
* Body weight ≥ 50 kg (110lbs) for males and ≥ 45 kg (99lbs) for females.
* Body mass index (BMI) within the range 18.5-35.0 kg/m2 inclusive.
* The subject has a diagnosis of RA according to the revised 1987 criteria of the American College of Rheumatology (ACR) (see Appendix 6).
* The subject must have DAS28 ≥ 4.2 (DAS28 calculated using ESR).
* The subject must have liver function (ALT, AST and total bilirubin) tests < 1.5 x ULN at screening.
* The subject must have ALP < 2 x ULN at screening.
* The subject must have normal serum folate levels at screening (folate supplements can be administered if required but this must be stable for 4 weeks prior to randomisation).
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.
* Signed and dated written informed consent prior to admission to the study.

Exclusion criteria:

* The subject has a three month prior history of regular alcohol consumption exceeding an average weekly intake of > 21 units (or an average daily intake of greater than 3 units) for males, or an average weekly intake of > 14 units (or an average daily intake of greater than 2 units) for females. 1 unit is equivalent to a half-pint (284mL) of beer/lager; 25mL measure of spirits or 125mL of wine; or a positive alcohol breath test at the screening visit.
* The subject has any history of liver disease.
* The subject has a positive Hepatitis B surface antigen or Hepatitis C antibody result within 3 months of the start of the study.
* The subject has a history of elevated liver function tests on more than one occasion (ALT, AST, and total bilirubin > 2 x ULN or ALP > 3 x ULN) in the past 7 months.
* The subject is currently receiving a biological anti-rheumatic therapy.
* The subject has failed more than one anti-TNFα biological therapy due to lack of efficacy.
* The subject received an anti-rheumatic biological therapy within 6 months (for i.v.

administered therapies with long half-lives e.g. infliximab) or 3 months (for subcutaneously administered therapies or iv administered therapies with short halflives e.g. adalimumab or etanercept) prior to randomisation.

* The subject has received rituximab.
* The subject is using oral prednisolone at doses > 10mg/day, methotrexate > 25 mg/week or sulphasalazine > 5g/day.
* The subject's DMARD dosing regimen has changed during the 4 weeks prior to randomisation.
* The subject's current DMARD regimen has changed significantly (i.e. likely to impact disease activity during the study period) within the 3 months prior to dosing e.g. addition of a DMARD, changes in dose of greater than 2.5mg for methotrexate.
* The subject has received leflunomide for less than 6 months prior to randomisation.
* The subject has failed more than 3 DMARDs.
* The subject's NSAIDs, COX-2 inhibitors or glucocorticoid dosing regimen changes at any time during four weeks prior to randomisation.
* The subject's statin dosing regimen has changed significantly during the 3 months prior to randomisation
* The subject has significant cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions that, in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as a participant in this trial.
* The subject has an acute infection or a history of repeated or chronic infections.
* The subject has a history of active tuberculosis.
* The subject has a history of malignancy, except for surgically cured basal cell carcinoma or females with cured cervical carcinoma (> 2 yrs prior).
* The subject has a history of HIV or other immunosuppressive disease.
* The subject has participated in a clinical trial within the 3 months prior to the study onset for non-biological therapy; or within 6 months of a biological therapy.
* The subject has Hb < 9 g/dL and platelet count < 150 000/mm3.
* The subject has a calculated creatinine clearance less than 60mL/min (subjects with a calculated creatinine clearance ≥ 50mL/min but < 60mL/min may still be included in consultation with the GSK medical monitor, but will not be eligible for the gadolinium enhancement MRI scans).
* The subject has uncontrolled diabetes or psoriasis.
* The subject has had a joint injection with glucocorticoid within the previous 4 weeks.
* The subject is pregnant or nursing.
* The subject is receiving medication which in the opinion of the investigator and/or GSK medical monitor, would interfere with study procedures, objectives or compromise subject safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Disease activity score based on 28 joint count (DAS28) at the end of the study. | at the end of the study.

SECONDARY OUTCOMES:
Adverse events, vitals signs, ECGs and clinical lab tests after 56 days. | after 56 days.
Plasma biomarkers after 56 days. | after 56 days
Population pharmacokinetics after 56 days | after 56 days
Gadolinium enhanced MRI scans after 56 days. | after 56 days.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- GSK Investigational Site, Bucharest, Romania
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Pertersburg
  - GSK Investigational Site, Yaroslavl
- Spain (3):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela

REFERENCES:
- [Derived] Yang S, Lukey P, Beerahee M, Hoke F. Population pharmacokinetics of losmapimod in healthy subjects and patients with rheumatoid arthritis and chronic obstructive pulmonary diseases. Clin Pharmacokinet. 2013 Mar;52(3):187-98. doi: 10.1007/s40262-012-0025-6. PMID 23254770